CLINICAL TRIAL: NCT01082822
Title: Periodontal Ligament Stem Cell Implantation in the Treatment of Periodontitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Professor Yan Jin, Research and Development Center for Tissue Engineering, Fourth Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEFMMU
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Periodontitis
Keywords: cell sheet PDLSC periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard of care (Sham Comparator): In the first step, the patient was periodontally treated until the inflammation was eliminated through control of bacterial biofilm and oral hygiene for about 6 months. Then the rigid fixed appliances were placed on the diseased teeth, reverse beveled open-flap surgery was performed in the buccal and palatal maxillary sides of the periodontitis-caught teeth to allow granulation tissue debridement and proper root preparation. The roots were completely scaled, and 17%EDTA was applied for 2 minutes to demineralize the root surfaces and bone wall defects, the flap was sutured.
  Interventions: Biological: cell sheet pellets and cell sheet fragment
- PDLSC cell sheet transplantion (Experimental): Periodontal ligament stem cell derived cell sheet or pellet with carrier such as Bioss was implanted into periodontal defect area at post surgical treatment.
  Interventions: Biological: cell sheet pellets and cell sheet fragment
- the bio-ss implantation (Experimental): implantation of Bioss at post surgical treatment
  Interventions: Biological: cell sheet pellets and cell sheet fragment

INTERVENTIONS:
Biological: cell sheet pellets and cell sheet fragment — the denuded root surface area was calculated to determine the size of the transplanted cell sheet in the of proportion of the 2cm X 2cm cell sheet to the 1cm X 1cm denuded area
  Other Names: cell sheet or pellet implantation

SUMMARY:
Cell sheet technique possess the properties of conserving the ECM, rich molecules and retaining cell vitality, and will promote the capacity of cell adhesion and proliferation. The stem cell based cell sheet therapy has been utilized in many fields and scored the satisfactory results. Periodontitis is a chronic disease which causes the destruction of the periodontal tissue and leads to the teeth loss in the end. The routine cell-based therapy to the periodontitis was confronted with many difficulties. In the investigators previous preclinical research, +the investigators fabricated periodontal ligament stem cell (PDLSC) pellets and cell sheet fragment and applied them in the periodontal defect area for tissue regeneration and periodontitis treatment. And the investigators carried out a comprehensive study of the PDLSC allograft. The host responses and implanted cell fates were recorded. After the scientific investigation of the preclinical study, the investigators designed the preliminary clinical trial of PDLSC cell sheet for the chronic periodontitis therapy in the aims to test the PDLSC fates and explore one ideal transplantation mode.

DETAILED DESCRIPTION:
our protocol mainly includes following steps:

1. select periodontitis patients :all patients were given the comprehensive examination on the oral condition including clinical examination, radiological evaluation and the immune system tests
2. select healthy donor teeth for PDLSC isolation and expansion.
3. fabricate the cell sheet and prepare the PDLSC cell sheet pellets and cell sheet fragment.
4. patients given the routine mechanical and chemical treatment for 4 weeks were randomized divided into 4 groups according to the visit time: i) the cell sheet fragment plus bio-ss transplantation; ii) the cell sheet pellets plus bioss transplantation; iii) the bio-ss transplantation and iv) the control.
5. all the operations were carried out as the routine GBR procedures.
6. the clinical, radiological examination and the changes of the immune system at the point of 1 day before and 4weeks, 12weeks, 24weeks and one year after the intervention were recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

1. adult chronic periodontitis
2. pathological lesion is stable after the routine mechanical and chemical treatment.
3. the local pathological lesion has the subbony defect
4. the oral heath was kept approved.
5. there are more 2 teeth with the continued lesion

Exclusion Criteria:

1. the age>50 year or < 40year
2. the patient has the genetic background of the periodontitis.
3. the bone destruction was larger than 2/3 of the root length.
4. the preclinical treatment was stable.
5. the severe systematic diseases.
6. the patients who can not cooperate with the whole the observation.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-11 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
The Plaque Index was mean score of each surface. Probing depth and Attachment loss are distance from the base of the sulcus and the cemento-enamel junction to the free gingival margin. bone loss | Sept. 2009

CONTACTS AND LOCATIONS:
Overall Officials: Yan Jin, PHD, Principal Investigator — Research and Development Center for Tissue Engineering, Fourth Military Medical University
Locations (1):
- Research and Develop Center for Tissue Engineering, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Yang Z, Jin F, Zhang X, Ma D, Han C, Huo N, Wang Y, Zhang Y, Lin Z, Jin Y. Tissue engineering of cementum/periodontal-ligament complex using a novel three-dimensional pellet cultivation system for human periodontal ligament stem cells. Tissue Eng Part C Methods. 2009 Dec;15(4):571-81. doi: 10.1089/ten.tec.2008.0561. PMID 19534606